CLINICAL TRIAL: NCT06441942
Title: Creation of a Prospective Multicenter Registry of Gender, Diversity and Inclusion (GEDI) in Phenotypic and Genetic Characterization of Acute Coronary Syndrome.
Brief Title: Prospective Multicenter Registry of Gender, Diversity and Inclusion (GEDI) of Women With Acute Coronary Syndrome
Acronym: ACS GEDI
Status: Not yet recruiting | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Collaborators: Federico II University (Other)
Responsible Party: Principal Investigator, Chieffo Alaide, Prof. M.D., IRCCS San Raffaele
Other Study IDs: PNRR-MCNT2-2023-12377431
Record Dates: First submitted 2024-05-29; First posted 2024-06-04 (Actual); Last update posted 2024-06-06 (Actual); Status verified 2024-06

CONDITIONS: Acute Coronary Syndrome; Gender; Genetic Predisposition
Keywords: ACS; GEDI; Genetic; DNA; mRNA; Proteomic; Metabolomic
MeSH Terms: conditions — Acute Coronary Syndrome; Coitus; Genetic Predisposition to Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Biospecimen Retention: Samples With DNA — DNA, mRNA, proteomic and metabolomic.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Case: Female patient presenting with ACS (age >/= 18)

SUMMARY:
Create a multicenter prospective registry that collects information from women affected by acute coronary syndrome (ACS). This registry aims to understand the diversity in the presentation of women with ACS. It proposes to conduct a thorough characterization of the women involved in the study through genetic, biochemical, and molecular analysis.This approach aims to identify any differences in the characteristics of women with ACS and to identify disease subtypes that may influence treatment options and clinical outcomes.

DETAILED DESCRIPTION:
Create a multicenter prospective registry that collects information from women affected by acute coronary syndrome (ACS) from a wide range of cultural and ethnic backgrounds distributed across various Italian regions. This registry aims to understand the diversity in the presentation of women with ACS in Italy, providing valuable data for a better understanding of the disease.

Additionally, it proposes to conduct a thorough characterization of the women involved in the study through genetic, biochemical, and molecular analysis. This analysis will be stratified by age and the etiology of coronary artery disease, distinguishing between obstructive and non-obstructive coronary artery disease.

Specific aims of this proposal are:

1. To create a multicenter prospective registry including women with ACS from a variety of cultural and ethnical backgrounds in different Italian regions
2. To deeply characterize women with ACS through clinical, imaging, genetic, biochemical, and molecular phenotyping stratifying for age, etiology (obstructive vs non-obstructive CAD) and diversity.
3. To assess socioeconomic status, health literacy and awareness of risk factors among enrolled patients.

ELIGIBILITY:
Inclusion Criteria:

* Women >/= 18 years with ACS (STEMI, NSTEMI or Unstable Angina).

Exclusion Criteria:

* age < 18 years and/or unwillingness to sign informed consent and/or unwillingness to make follow-up visits

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female patient >/= 18
Study Population: The study will include female patients presenting with ACS (according to ESC guidelines)
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2025-07-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Multicentric Registry | 12 months of follow-up
  The aim will be to create a prospective multicenter registry of gender, diversity and inclusion (GEDI) of women with Acute Coronary Syndrome

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS San Raffaele Hospital, Milan, Italy Milan, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Weiss AM. Cardiovascular disease in women. Prim Care. 2009 Mar;36(1):73-102, viii. doi: 10.1016/j.pop.2008.10.012. PMID 19231603
- [Background] Vogel B, Acevedo M, Appelman Y, Bairey Merz CN, Chieffo A, Figtree GA, Guerrero M, Kunadian V, Lam CSP, Maas AHEM, Mihailidou AS, Olszanecka A, Poole JE, Saldarriaga C, Saw J, Zuhlke L, Mehran R. The Lancet women and cardiovascular disease Commission: reducing the global burden by 2030. Lancet. 2021 Jun 19;397(10292):2385-2438. doi: 10.1016/S0140-6736(21)00684-X. Epub 2021 May 16. PMID 34010613
- [Background] Graham G. Acute Coronary Syndromes in Women: Recent Treatment Trends and Outcomes. Clin Med Insights Cardiol. 2016 Feb 8;10:1-10. doi: 10.4137/CMC.S37145. eCollection 2016. PMID 26884685
- [Background] Vaccarino V, Parsons L, Every NR, Barron HV, Krumholz HM. Sex-based differences in early mortality after myocardial infarction. National Registry of Myocardial Infarction 2 Participants. N Engl J Med. 1999 Jul 22;341(4):217-25. doi: 10.1056/NEJM199907223410401. PMID 10413733
- [Background] Udell JA, Fonarow GC, Maddox TM, Cannon CP, Frank Peacock W, Laskey WK, Grau-Sepulveda MV, Smith EE, Hernandez AF, Peterson ED, Bhatt DL; Get With The Guidelines Steering Committee and Investigators. Sustained sex-based treatment differences in acute coronary syndrome care: Insights from the American Heart Association Get With The Guidelines Coronary Artery Disease Registry. Clin Cardiol. 2018 Jun;41(6):758-768. doi: 10.1002/clc.22938. Epub 2018 May 11. PMID 29521450
- [Background] Bavishi C, Bangalore S, Patel D, Chatterjee S, Trivedi V, Tamis-Holland JE. Short and long-term mortality in women and men undergoing primary angioplasty: A comprehensive meta-analysis. Int J Cardiol. 2015 Nov 1;198:123-30. doi: 10.1016/j.ijcard.2015.07.001. Epub 2015 Jul 4. PMID 26163903
- [Background] Renda G, Patti G, Lang IM, Siller-Matula JM, Hylek EM, Ambrosio G, Haas S, De Caterina R; Working Group on Thrombosis of the Italian Society of Cardiology. Thrombotic and hemorrhagic burden in women: Gender-related issues in the response to antithrombotic therapies. Int J Cardiol. 2019 Jul 1;286:198-207. doi: 10.1016/j.ijcard.2019.02.004. Epub 2019 Feb 8. PMID 30777407
- [Background] Smilowitz NR, Mahajan AM, Roe MT, Hellkamp AS, Chiswell K, Gulati M, Reynolds HR. Mortality of Myocardial Infarction by Sex, Age, and Obstructive Coronary Artery Disease Status in the ACTION Registry-GWTG (Acute Coronary Treatment and Intervention Outcomes Network Registry-Get With the Guidelines). Circ Cardiovasc Qual Outcomes. 2017 Dec;10(12):e003443. doi: 10.1161/CIRCOUTCOMES.116.003443. PMID 29246884
- [Background] Wechkunanukul K, Grantham H, Damarell R, Clark RA. The association between ethnicity and delay in seeking medical care for chest pain: a systematic review. JBI Database System Rev Implement Rep. 2016 Jul;14(7):208-35. doi: 10.11124/JBISRIR-2016-003012. PMID 27532797
- [Background] Bonaccorsi G, Grazzini M, Pieri L, Santomauro F, Ciancio M, Lorini C. Assessment of Health Literacy and validation of single-item literacy screener (SILS) in a sample of Italian people. Ann Ist Super Sanita. 2017 Jul-Sep;53(3):205-212. doi: 10.4415/ANN_17_03_05. PMID 28956799
- [Background] Parker RM, Baker DW, Williams MV, Nurss JR. The test of functional health literacy in adults: a new instrument for measuring patients' literacy skills. J Gen Intern Med. 1995 Oct;10(10):537-41. doi: 10.1007/BF02640361. PMID 8576769
- [Background] Byrne RA, Rossello X, Coughlan JJ, Barbato E, Berry C, Chieffo A, Claeys MJ, Dan GA, Dweck MR, Galbraith M, Gilard M, Hinterbuchner L, Jankowska EA, Juni P, Kimura T, Kunadian V, Leosdottir M, Lorusso R, Pedretti RFE, Rigopoulos AG, Rubini Gimenez M, Thiele H, Vranckx P, Wassmann S, Wenger NK, Ibanez B; ESC Scientific Document Group. 2023 ESC Guidelines for the management of acute coronary syndromes. Eur Heart J. 2023 Oct 12;44(38):3720-3826. doi: 10.1093/eurheartj/ehad191. No abstract available. PMID 37622654
- [Background] Agewall S, Beltrame JF, Reynolds HR, Niessner A, Rosano G, Caforio AL, De Caterina R, Zimarino M, Roffi M, Kjeldsen K, Atar D, Kaski JC, Sechtem U, Tornvall P; WG on Cardiovascular Pharmacotherapy. ESC working group position paper on myocardial infarction with non-obstructive coronary arteries. Eur Heart J. 2017 Jan 14;38(3):143-153. doi: 10.1093/eurheartj/ehw149. No abstract available. PMID 28158518
- [Background] Collet JP, Thiele H, Barbato E, Barthelemy O, Bauersachs J, Bhatt DL, Dendale P, Dorobantu M, Edvardsen T, Folliguet T, Gale CP, Gilard M, Jobs A, Juni P, Lambrinou E, Lewis BS, Mehilli J, Meliga E, Merkely B, Mueller C, Roffi M, Rutten FH, Sibbing D, Siontis GCM; ESC Scientific Document Group. 2020 ESC Guidelines for the management of acute coronary syndromes in patients presenting without persistent ST-segment elevation. Eur Heart J. 2021 Apr 7;42(14):1289-1367. doi: 10.1093/eurheartj/ehaa575. No abstract available. PMID 32860058
- [Background] Sousa-Uva M, Neumann FJ, Ahlsson A, Alfonso F, Banning AP, Benedetto U, Byrne RA, Collet JP, Falk V, Head SJ, Juni P, Kastrati A, Koller A, Kristensen SD, Niebauer J, Richter DJ, Seferovic PM, Sibbing D, Stefanini GG, Windecker S, Yadav R, Zembala MO; ESC Scientific Document Group. 2018 ESC/EACTS Guidelines on myocardial revascularization. Eur J Cardiothorac Surg. 2019 Jan 1;55(1):4-90. doi: 10.1093/ejcts/ezy289. No abstract available. PMID 30165632
- See also: Related Info — https://www.un.org/sustainabledevelopment/health/
- See also: Related Info — https://euroqol.org/information-and-support/euroqol-instruments/eq-5d-5l/